CLINICAL TRIAL: NCT04493606
Title: Implementation of the ProACTIVE Toolkit in the Hospital and Community Setting to Improve Physical Activity Among People With Spinal Cord Injury
Brief Title: Implementation of the ProACTIVE Toolkit in the Hospital and Community Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Rick Hansen Institute (Other)
Responsible Party: Principal Investigator, Kathleen Martin Ginis, Professor, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ProACTIVE Implementation
Record Dates: First submitted 2020-07-10; First posted 2020-07-30 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Patients (Experimental): SCI patients receiving the physical activity coaching (Objective 1)
  Interventions: Other: SCI ProACTIVE Coaching (objective 1)
- Intervention- Interventionists (Experimental): Interventionists receiving physical activity coaching training (Objective 2)
  Interventions: Behavioral: Implementation Intervention (objective 2)

INTERVENTIONS:
Other: SCI ProACTIVE Coaching (objective 1) — Peer coaches will conduct an assessment to understand patient's readiness, goals, barriers, preferences, and access to physical activity resources and mutually select tailored physical activity-enhancing strategies based on the assessment. These strategies include education (SCI exercise guidelines, safety, benefits, basics of physical activity, behaviour change techniques) and referral to appropriate peers, programs, and organizations. Goals will be based on the SCI Fitness Guidelines (targeting a goal of 20min of moderate to vigorous intensity aerobic exercise + 3 sets of strength training exercises for each major functioning muscle group at a moderate to vigorous intensity each 2x/week) and if ready, the Canadian SCI Physical Activity Guidelines (30 min 3x/week of moderate to vigorous intensity aerobic exercise + strength training 2x/ week). Ten 15-minute, video-conference or telephone sessions will be scheduled in accordance with patient needs and readiness with the peer coaches.
  Arms: Intervention Patients
Behavioral: Implementation Intervention (objective 2) — A training on how to deliver the ProACTIVE intervention will be delivered. Day 1 training will include an overview of the intervention, demonstration of the delivery of the intervention, and behavioural practice. Interventionists will practice delivering the intervention and record issues or questions to bring to the day 2 training. Day 2 training will include a refresher on intervention content, barriers identified during in-clinic/community practice will be addressed, and further behavioural practice with volunteer clients with additional feedback provided.
  The trainer (Dr. Jasmin Ma) will provide monitoring and feedback during the first two months of implementation. Community of practice meetings will be held as needed to discuss challenges and facilitators to implementation. Feedback provided during community of practice meetings will be collected and used for iterative quality improvement of the intervention approaches.
  Arms: Intervention- Interventionists

SUMMARY:
There is a significant drop in physical activity among people with spinal cord injury in the months following discharge from rehabilitation. The ProACTIVE toolkit is a guide to promote physical activity to clients with spinal cord injury that has demonstrated potential to help address this sensitive time frame for physical inactivity. The toolkit was co- developed with 300 physiotherapists, community members with spinal cord injury, and university researchers and has been shown to improve physical activity and fitness in this population. Physiotherapists will refer clients to peer coaches with spinal cord injury who will implement the toolkit. The investigators will assess how well the toolkit is used and its effectiveness to improve physical activity levels.

DETAILED DESCRIPTION:
Purpose 1 (arms 1 and 2): To evaluate the effect of referral to peer-led coaching, guided by the ProACTIVE SCI intervention, on physical activity behaviour, health, and quality of life outcomes among people with SCI.

Procedure overview: Participants will complete survey measures (~45 minutes) at baseline/discharge, 2 months, 6 months post discharge, and 1-year follow-up. Participants will also complete a semi-structured interview to assess satisfaction with the intervention at 6 months. Participants in the intervention group will receive an initial assessment (~1 hour) and 10 physical activity coaching sessions (~15 minutes each). A total time commitment of ~6.5 hours is expected over one year.

Design: For pragmatic and ethical reasons, single-group, repeated measures design will be used where interested participants will receive the intervention.

Procedure: Patients who are interested in participating will be enrolled in the intervention and will receive the ProACTIVE SCI intervention coaching. Patients who are not interested in participating will be re-contacted before discharge and/or at 3 months post-discharge to gauge interest. For those who consent during their hospital stay, a two-page quick-sheet will be filled out at discharge to record any physical activity coaching information collected during their hospital stay as part of usual care. (Please see Section 9 for the "GF Strong inpatient/ form" and "GF Strong outpatient form" that is currently used in practice). The quick-sheet and any exercise prescriptions developed will be transferred to the SCI BC peers. If possible, SCI BC peers will contact the client in-person or over video-conference before discharge to begin coaching, otherwise SCI BC peers will contact the patient to begin coaching sessions in the community post-discharge. SCI BC peers will carry out the physical activity coaching sessions guided by the ProACTIVE SCI intervention with the exception that exercise prescriptions cannot be made by the peers. If exercise prescriptions are needed, referral to an adapted personal trainer in the community will be made. Coaching sessions will be provided either in-person, using video teleconferencing technology or telephone if needed. Ten 15-minute sessions will be scheduled in accordance with patient needs and readiness, however, as a general structure, one coaching session will be provided each month for months 1-3, two coaching sessions per month in months 4-6, with a follow-up before one year. The peer coaches will make up to 5 attempts to reschedule a missed coaching session.

Sample size estimate: Based on feasibility estimates calculated using number of patients admitted yearly to GF Strong (n=100), an estimated 70% discharged to home (n=70; remaining 30% discharged to long-term care or other), approximately 55% of patients willing to consent over the 3 month follow-up period, and a 20% dropout estimate (based on previous experience in conducting studies in this population) an estimated n=30 individuals will be recruited to the intervention group (see Figure 2).

To ensure the sample size based on feasibility is adequately powered to detect an effect on physical activity, the investigators conducted a power calculation based on a previous randomized controlled trial in the in-patient setting with individuals with spinal cord injury. Physiotherapists delivered a bi-weekly behavioural coaching intervention to 39 individuals with SCI and physical activity was assessed at baseline, discharge, 6-months, and one-year post-discharge. A large-sized effect was observed at 6 months (d=0.89) for self-reported physical activity. Given the quasi-experimental design, the investigators are powering for a more modest between groups difference (d = .75). Eight participants/condition (N = 16) are needed to yield a significant effect of this magnitude in a repeated measures ANOVA, with β = .80 and α = .05. Thus, the feasibility-based projected sample size is adequate to detect a significant effect of the intervention on physical activity in this context.

Statistical Analysis: One-way repeated measures ANOVA

Purpose 2 (arm 3): Evaluate, understand, and document the implementation process of physiotherapists and peers with SCI delivering the ProACTIVE SCI intervention

Procedure overview: Clinicians and SCI BC Peers will receive a two-day training (2 hours each day) on how to deliver the ProACTIVE intervention. Clinicians and SCI BC Peers will be supported with monitoring and feedback for the first two months of delivering the intervention to clients and community of practice meetings as needed. 20-minute surveys will be administered before and immediately after training, as well as at 2 months and 6 months after starting implementation. One-hour semi-structured interviews will be conducted at 6 months. A total time commitment of ~18.5 hours is expected over one year for the clinicians. SCI BC Peers will deliver 10x15 minute coaching sessions to ~ 10 participants each for a total time commitment of 43.5 hours over one year.

Design: Within-subject, repeated measures.

Participants: As the aim of this project is to deliver the intervention using a pragmatic approach, volunteer physiotherapists from GF Strong and SCI BC peer coordinators who are interested in delivering the ProACTIVE SCI intervention will be included in this objective.

Sample size estimate: The study is powered to detect a significant within-subject effect over time on the theoretical domains framework (TDF) measures. A previous evaluation of the ProACTIVE implementation training amongst physiotherapists, when using within subject pre-post analyses, demonstrated a very large effect size across TDF outcomes (f=.867). A minimum of five participants are needed to yield a significant effect of this magnitude in a within-subject, repeated measures ANOVA (4 time points), with β = .80, α = .05, and a conservative 0.25 correlation among repeated measures.

Statistical Analysis: One-way repeated measure ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* traumatic or non-traumatic spinal cord injury
* do not require ventilatory assistance, and
* have no medical contraindications to exercise identified by the care team

Exclusion Criteria:

* Uncontrolled symptoms of cardiovascular disease or cardiopulmonary problems/disease.
* Active Stage 3 or 4 pressure ulcer (based on the National Pressure Ulcer Advisory Panel classification)
* Any unstable medical/psychiatric condition or substance abuse disorder that is likely to affect their ability to complete this study.- Any cognitive dysfunction or language barrier that would prevent subjects from following English instructions.
* Participants may be excluded at the discretion of the principal investigator due to other, unforeseen, safety issues.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Leisure Time Physical Activity at 1 month, 6 months, and 1 year | Baseline, 1 month, 6 month, 1 year
  Measures include the Leisure Time Physical Activity Questionnaire for People with SCI, which is a self-report measure that assesses minutes of mild, moderate, and vigorous intensity leisure time physical activity (i.e., activity that requires physical exertion and that one chooses to do in their free time) that is broken down into strength training and aerobic activity performed over the past seven days. Lower scores reflect less participation in leisure time physical activity. Support for the Leisure Time Physical Activity Questionnaire's criterion validity and test-retest reliability has been previously demonstrated in a sample of 103 men and women with SCI.

SECONDARY OUTCOMES:
Psychosocial predictors of physical activity | Baseline, 1 month, 6 month, 1 year
  Psychosocial predictors of physical activity will be assessed using a survey based on the Health Action Process Approach (HAPA) model. Measures of the HAPA constructs are drawn from existing measures and previous SCI studies where possible. All items are assessed on a 7-point Likert scale ranging from 1='strongly disagree' to 7='strongly agree'. The survey will be recorded either electronically or with pen and paper depending on the respondent's preference. Survey will take approximately 25 minutes to complete, and will assess constructs related to exercise such as perceived risks, self- efficacy, planning, and social support. The demographics questionnaire will also be administered with this measure.

OTHER OUTCOMES:
Determinants of implementation behaviour for interventionists | Baseline, 1 month, 6 month, 1 year
  Intervention delivers will be asked to complete an online implementation questionnaire guided by the theoretical domains framework to assess factors that affect delivery of the intervention. The questionnaire consists of 40 questions; eight questions on a 6-point Likert scale where higher scores indicated greater implementation of the toolkit, and 32 questions on an 8-point Likert scale where higher scores indicate greater agreement with factors associated with the implementation.
Semi-structured interviews- interventionists | 6 months
  Sixty-minute individual interviews will be conducted. Semi-structured interviews will explore interventionist experiences, needs, and factors (barriers and facilitators) that affect physical activity coaching behaviour guided by the ProACTIVE SCI intervention. Interviews will be recorded and transcribed verbatim
Semi-structured interviews- Patients | 1 year
  Sixty-minute individual interviews will be conducted. Semi-structured interviews will be conducted over the phone or video conference. Semi-structured interviews will explore the impacts of the intervention on physical and mental health, use of healthcare services, quality of life, and function, as well as participants' satisfaction and future recommendations for the coaching intervention. Interviews will be recorded and transcribed verbatim.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Martin Ginis, PhD, Principal Investigator — University of British Columbia
Locations (1):
- GF Strong Rehabilitation Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bandura, A. (1997). Self-efficacy: The Exercise of Control. New York: W.H. Freeman & Co.
- [Background] Brawley LR, Arbour-Nicitopoulos KP, Martin Ginis KA. Developing physical activity interventions for adults with spinal cord injury. Part 3: a pilot feasibility study of an intervention to increase self-managed physical activity. Rehabil Psychol. 2013 Aug;58(3):316-21. doi: 10.1037/a0032814. PMID 23978087
- [Background] Caspersen CJ, Powell KE, Christenson GM. Physical activity, exercise, and physical fitness: definitions and distinctions for health-related research. Public Health Rep. 1985 Mar-Apr;100(2):126-31. PMID 3920711
- [Background] Cowan RE, Nash MS, Anderson KD. Exercise participation barrier prevalence and association with exercise participation status in individuals with spinal cord injury. Spinal Cord. 2013 Jan;51(1):27-32. doi: 10.1038/sc.2012.53. Epub 2012 May 15. PMID 22584283
- [Background] Ma JK, Cheifetz O, Todd KR, Chebaro C, Phang SH, Shaw RB, Whaley KJ, Martin Ginis KA. Co-development of a physiotherapist-delivered physical activity intervention for adults with spinal cord injury. Spinal Cord. 2020 Jul;58(7):778-786. doi: 10.1038/s41393-020-0422-x. Epub 2020 Jan 22. PMID 31969687
- [Background] Ginis KA, Hicks AL, Latimer AE, Warburton DE, Bourne C, Ditor DS, Goodwin DL, Hayes KC, McCartney N, McIlraith A, Pomerleau P, Smith K, Stone JA, Wolfe DL. The development of evidence-informed physical activity guidelines for adults with spinal cord injury. Spinal Cord. 2011 Nov;49(11):1088-96. doi: 10.1038/sc.2011.63. Epub 2011 Jun 7. PMID 21647164
- [Background] Martin Ginis KA, Phang SH, Latimer AE, Arbour-Nicitopoulos KP. Reliability and validity tests of the leisure time physical activity questionnaire for people with spinal cord injury. Arch Phys Med Rehabil. 2012 Apr;93(4):677-82. doi: 10.1016/j.apmr.2011.11.005. Epub 2012 Feb 13. PMID 22336103
- [Background] Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader PR. The development of scales to measure social support for diet and exercise behaviors. Prev Med. 1987 Nov;16(6):825-36. doi: 10.1016/0091-7435(87)90022-3. PMID 3432232
- [Background] Scholz, U., Sniehotta, F. F., & Schwarzer, R. (2005). Predicting physical exercise in cardiac rehabilitation: The role of phase-specific self-efficacy beliefs. Journal of Sport and Exercise Psychology, 27(2), 135-151
- [Background] Schwarzer R, Lippke S, Luszczynska A. Mechanisms of health behavior change in persons with chronic illness or disability: the Health Action Process Approach (HAPA). Rehabil Psychol. 2011 Aug;56(3):161-70. doi: 10.1037/a0024509. PMID 21767036
- [Background] Sniehotta, F. F., Scholz, U., & Schwarzer, R. (2005). Bridging the intention-behaviour gap: Planning, self-efficacy, and action control in the adoption and maintenance of physical exercise. Psychology & Health, 20(2), 143-160. https://doi.org/10.1080/08870440512331317670
- [Derived] Ma JK, Walden K, McBride CB, Le Cornu Levett C, Colistro R, Plashkes T, Thorson T, Shu H, Martin Ginis KA. Implementation of the spinal cord injury exercise guidelines in the hospital and community settings: Protocol for a type II hybrid trial. Spinal Cord. 2022 Jan;60(1):53-57. doi: 10.1038/s41393-021-00685-7. Epub 2021 Aug 10. PMID 34376809